CLINICAL TRIAL: NCT04869540
Title: Improving Transition Outcomes for Youth With Autism Spectrum Disorder From Within a Medicaid Accountable Care Organization
Brief Title: Improving Transition Outcomes for Youth With ASD in a Medicaid Accountable Care Organization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Investigator left the institution and the study was not implemented.
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-41693; 5K18MH120457 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Transition-aged youth (TAY); Medicaid ACO; Got Transition toolkit; Problem solving education (PSE)
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Families randomized to this arm will receive the usual care by providers trained in the 'Got Transition' toolkit and that have access to web-based transition resources.
  Interventions: Other: Usual care; Other: 'Got Transition' toolkit and resources
- Usual care + PSE (Experimental): Families randomized to this arm will receive the usual care by providers trained in the 'Got Transition' toolkit and that have access to web-based transition resources and will also receive a family-based problem solving eduction (PSE) intervention.
  Interventions: Other: Usual care; Other: 'Got Transition' toolkit and resources; Behavioral: PSE intervention

INTERVENTIONS:
Other: Usual care — Evidence based care for transition-aged youth (TAY) with ASD.
Other: 'Got Transition' toolkit and resources — Providers will be trained in the 'Got Transition' toolkit (the systems level component of the intervention) and have access to web-based transition resources.
Behavioral: PSE intervention — A family-based problem solving education (PSE) intervention.
  Arms: Usual care + PSE

SUMMARY:
Despite an increasing number of children with Autism Spectrum Disorder (ASD), fragmentation across child and adult service systems results in poor education, employment and health outcomes for transition-aged youth (TAY). The investigators will develop a transition intervention embedded in a series of systems-level strategies currently being deployed in a large Medicaid Accountable Care Organization (ACO). The investigators will conduct a randomized pilot study of 40 families of TAY with ASD. All families will receive care by providers trained in the Got Transition toolkit (the systems level component of the intervention) and have access to web-based transition resources. Families in the 'intervention refinement' arm will also receive a family-based problem solving education (PSE) intervention.

DETAILED DESCRIPTION:
This is a randomized pilot study of 40 families of TAY with ASD. Families will be randomly allocated to study arms - not for the purpose of maximizing internal validity; but rather, to allow us to refine recruitment techniques that maximize the acceptability of randomization. Twenty families in the 'intervention refinement' arm will receive a PSE-based intervention; among this group, the model will be refined in real time - based on both experience delivering the intervention and ongoing qualitative data collection. Refinement arm participants will receive a PSE prototype based on prior initial adaptations.

Each pilot family will also be asked to participate in a semi-structured interview. The interviews will be conducted after families have experienced at least 3 PSE sessions and use their data to further refine the model and develop hypotheses concerning testable intervention targets.

Among 20 families in a control-like 'parameter estimation' arm, empiric estimates will be obtained of study parameters key to the design of a future trial. All families in this arm will receive care from providers trained in the Got Transition toolkit, and will have access to web-based resources for creating a young adult vision statement and for accessing multiple service sectors. Participants will be tracked over six-months. Consistent with pilot methods, the analysis will not emphasize comparisons across study arms

ELIGIBILITY:
Caregivers 18+ and transition aged youth with autism ages 14-20

Inclusion Criteria:

* Speak English or Spanish

Exclusion Criteria:

* Foster families
* Families in which a parent has either serious mental illness or limited cognitive capacity

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT) ASD | Baseline
  The PEDI-CAT ASD is a parent report measure that assesses abilities in three functional domains: Daily Activities, Mobility, and Social/Cognitive. A separate Responsibility domain measures the extent to which the caregiver or child takes responsibility for managing complex life tasks that enable independent living in the areas of Organization & Planning, Taking Care of Daily Needs, Health Management, and Staying Safe. The PEDI-CAT is valid up to age 21 and is specific to youth with ASD. Normative standard scores (provided as age percentiles and T scores) and Scaled Scores are available for 59 age groups. Typically, T-scores between 30 and 70 (i.e. mean ± 2 standard deviations) are considered within the expected range for age.
6 months PEDI-CAT ASD | 6 months
  The PEDI-CAT ASD is a parent report measure that assesses abilities in three functional domains: Daily Activities, Mobility, and Social/Cognitive. A separate Responsibility domain measures the extent to which the caregiver or child takes responsibility for managing complex life tasks that enable independent living in the areas of Organization & Planning, Taking Care of Daily Needs, Health Management, and Staying Safe. The PEDI-CAT is valid up to age 21 and is specific to youth with ASD. Normative standard scores (provided as age percentiles and T scores) and Scaled Scores are available for 59 age groups. Typically, T-scores between 30 and 70 (i.e. mean ± 2 standard deviations) are considered within the expected range for age.

SECONDARY OUTCOMES:
Social skills | baseline
  The 65 item Social Responsiveness Scale-2 assesses social impairment associated with ASD. Results are reported as T-scores for 5 treatment subscales: Social Awareness- 8 items to measure the ability to recognize social cues of others; Social Cognition- 12 items that addresses interpretation of social behavior; Social Communication- 22 items to assess reciprocal communication in social situations; Social Motivation- 11 items that assesses an individual's motivation to participate in social interactions; Restricted Interests & Repetitive Behavior- a 12 items that measures stereotypes and circumscribed interests; and the total score. T-scores of >76 are severe suggesting clinically significant deficits in social functioning that interfere with interactions with others. Scores 66-75 are moderate, signaling some clinically significant social deficits. T-scores of 60-65 indicate mild to moderate deficiencies in social behavior. T-scores < 60 indicate few social difficulties.
Cognition | baseline
  The Wechsler Abbreviated Scale of Intelligence (WASI) is a validated, time-efficient which will be used to measure of cognition/cognitive ability. The average score is fixed at 100, with approximately two-thirds of all scores falling somewhere between 85 and 115. HIgher scores are correlated with higher cognition.
Parent Functioning and Depressive Symptoms assessed by SAS-SR | baseline
  The Social Adjustment Scale Self-Report (SAS-SR) examines functioning in six areas, including role as parent. Raw scores are converted to gender-based standard scores (including T-scores and percentiles), with higher scores indicating higher levels of impairment (i.e., lower levels of social adjustment).
Parent Functioning and Depressive Symptoms assessed by QIDS | baseline
  The 16 item Quick Inventory of Depressive Symptoms (QIDS) is valid and reliable measure of depressive symptoms. Total QIDS scores range from 0 to 27 with scores of 5 or lower indicative of no depression, scores from 6 to 10 indicating mild depression, 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Family Empowerment | baseline
  The Family Empowerment Scale is a validated 34-item instrument developed to measure empowerment in families with children who have emotional, behavioral, or mental disorders. Responses are from 1=not at all to 5= Very true with a range of scores form 34 to 170. Higher scores are correlated with more family empowerment.
Perceived parental stress | baseline
  The 10 item perceived stress scale (PSS) will be used to assess parental stress. It includes domains in unpredictability, lack of control, burden overload, and stressful circumstances. 10 scores are obtained by reversing the scores on the four positive items. Scores around 13 are considered average. HIgher scores are correlated with more stress.
Parental stress | baseline
  The 13 item Autism Parenting Stress Index (APSI) will be used to assess how much stress parents are experiencing and what factors are causing this stress. The Items fall into three categories: the core social disability, difficult-to-manage behaviour, and physical issues. Items are rated as being 'Not stressful', 'Sometimes creates stress', 'Often creates stress', 'Very stressful on a daily basis', to 'So stressful that sometimes we feel we cannot cope.' Scores can rage form 0 to 65 and higher scores are correlated with more stress.
Perceived youth stress | baseline
  The 10 item perceived stress scale (PSS) will be used to assess youth stress. It includes domains in unpredictability, lack of control, burden overload, and stressful circumstances. 10 scores are obtained by reversing the scores on the four positive items. Scores around 13 are considered average. HIgher scores are correlated with more stress.
Parental coping strategies | baseline
  The 26 item Coping Self-Efficacy Scale will be used to measure the parent's ability to cope with life challenges in three domains: problem-focused coping, unpleasant thoughts, and getting support from others. Respondents are asked asked to rate on an 11-point scale the extent to which they believe they could perform behaviors important to adaptive coping. Anchor points on the scale are 0 ('cannot do at all'), 5 ('moderately certain can do') and 10 ('certain can do'). Higher scores are correlated with better coping strategies.
Youth coping strategies | baseline
  The 26 item Coping Self-Efficacy Scale will be used to measure the youth's ability to cope with life challenges in three domains: problem-focused coping, unpleasant thoughts, and getting support from others. Respondents are asked asked to rate on an 11-point scale the extent to which they believe they could perform behaviors important to adaptive coping. Anchor points on the scale are 0 ('cannot do at all'), 5 ('moderately certain can do') and 10 ('certain can do'). Higher scores are correlated with better coping strategies.
Vocational and Educational Activities | 6 months
  The Vocational Index is a valid index of vocational and educational outcomes for youth and young adults with ASD. It has 11 categories coded on a 9-point scale, ranging from competitive employment and/or postsecondary educational program to no vocational/educational activities. HIgher scores are correlated with greater vocational and educational activities.
Health Care Transition Readiness and Family Perception of Health Care Integration using TRAQ | 6 months
  The Transition Readiness Assessment Questionnaire (TRAQ) is a 20-item, 5-factor structure validated scale that assesses youths' ability to make appointments, understand medications and develop other transition skill. Answers are reported on a 1 to 5 scale based on the Stages of Change Model ranging from "I do not need to do this" to "I always do this when I need to." HIgher scores are correlated with greater transition readiness.
Health Care Transition Readiness and Family Perception of Health Care Integration using the Pediatric Integrated Care Survey (PICS) | 6 months
  PICS is a 48 item survey designed to assess families' experience of health care integration. A composite score is derived based on the response and higher scores are correlated with greater transition readiness and health care integration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD MPH, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No